CLINICAL TRIAL: NCT03461653
Title: Efficacy of Medical Abortion Through Telemedicine Versus Standard Provision - a Randomised Controlled Non-inferiority Trial
Brief Title: Telemedicin Counselling for Medical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: wow2018
Record Dates: First submitted 2018-02-28; First posted 2018-03-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Medical Abortion Counselling

STUDY DESIGN:
Intervention Model Description: Randomised trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine counselling (Other): intervention group Women who will receive telemedicine counselling
  Interventions: Other: Telemedicine counselling
- Standard care (No Intervention): Women who will receive standard face-to-face counselling

INTERVENTIONS:
Other: Telemedicine counselling — women on web counselling
  Arms: Telemedicine counselling

SUMMARY:
The guidance on Safe abortion technology by the World Health Organization (WHO 2012) suggests the evaluation of internet provision and telemedicine, as further alternative service delivery channels of safe abortion, as a subject for future research (WHO 2012) Our studies have shown that telemedicine and provision of medical abortion through wow is safe, acceptable and with outcomes similar to medical abortion provided traditionally following face-to-face counselling. Furthermore, recently home self-assessment of the abortion outcome through a low sensitivity U-hCg test was shown to be highly acceptable to women. To evaluate whether counselling through telemedicine is non-inferior to face-to face counselling a RCT will be conducted including women who chose medical abortion up to 63 days of gestation with home administration of misoprostol and self assessment of the outcome. The results of this study could be of major importance to increase access to safe and acceptable abortion services.

ELIGIBILITY:
Inclusion Criteria:

* requesting termination of pregnancy by means of mifepristone followed by home administration of misoprostol at < /=63 days of gestation, no contraindication to medical abortion and self administration of misoprostol at home, and who have given their informed consent

Exclusion Criteria:

* women who do not want home administration of misoprostol, women who are unable to communicate in Swedish, or English, and women with symptoms and signs of ectopic pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1598 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of women with complete abortion | 30 days of abortion treatment
  Efficacy of medical abortion defined as complete abortion without ongoing intrauterine pregnancy or surgical intervention for incomplete abortion within 30 days of the abortion treatment.Reported by the patient in the follow up questionnaire and by assessment of patient records

SECONDARY OUTCOMES:
Rate of reported complications that require additional treatment. | 30 days
  complications defined as; infection, bleeding Reported at follow up or
Proportions of women who would chose the same mode of provision in case of a future medical abortion | 30 days
  satisfaction with mode of counselling. Follow up questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2000-05-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT03461653/Prot_SAP_000.pdf